CLINICAL TRIAL: NCT05867446
Title: The Effect of Education Given to Hemodialysis Patients With Pecha Kuka Method on Attitude Towards Diet Therapy and Compliance With Fluid Restriction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, gülcan bahcecioğlu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/ 04- 12
Record Dates: First submitted 2023-04-12; First posted 2023-05-22 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Hemodialysis Patients
Keywords: diet; liquid; patients; nurse

STUDY DESIGN:
Intervention Model Description: pecha kucha training
Who Masked: Participant
Masking Description: Single (Participant) To Diet Therapy Attitude Towards Fluid Restriction Compliance
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: (Experimental): pecha kucha will be practiced
  Interventions: Behavioral: pecha kucha
- control (No Intervention): Routine maintenance will be applied.

INTERVENTIONS:
Behavioral: pecha kucha — pecha kucha training
  Arms: Experimental:

SUMMARY:
Hemodialysis complex treatment regimen includes fluid and diet management. In this context, it is recommended that patients choose foods with low sodium, potassium and phosphorus content, maintain adequate protein intake, and regulate their daily fluid intake not exceeding 1-2 liters. In maintaining the health of hemodialysis patients; It is very important that they comply with the treatment program, diet and fluid restrictions. As the life expectancy increases, the time spent with chronic disease also increases, and both the patient himself and his relatives living in the same house are faced with this chronic disease and accompanying stress factors for a longer period of time, making it difficult for them to adapt to the progression of the disease.

Pecha Kucha (PK), meaning "chat voice" or "chat" in Japanese, refers to a well-crafted, fast and concise presentation format. In a PK presentation, each presenter is only allowed to show 20 PowerPoint slides for 20 seconds each on a timer. When the literature was examined, no study was found that evaluated the effect of the education given to hemodialysis patients with the Pecha Kuka method on the attitude towards diet therapy and compliance with fluid restriction. In addition, it is thought that this short and concise education method will contribute to a better understanding of the attitudes of patients receiving hemodialysis treatment towards diet therapy and their compliance with fluid restriction, thus providing important data for future studies.

DETAILED DESCRIPTION:
Diet is one of the most important elements of HD treatment. Kidney disease can be slowed down with diet. There are important issues in the diet of individuals receiving HD treatment. Adequate energy consumption comes first. Individuals receiving HD treatment must meet the energy requirements needed to maintain their health, as well as perform their metabolic functions. Adequate protein intake is one of the important issues in the diet in patients receiving HD treatment. Compliance with disease treatment; it is briefly defined as "individual compliance with medical treatment and health recommendations". During the period of hemodialysis treatment, one of the areas where individuals have difficulty in adapting is diet and fluid restriction. Because the disease and HD treatment directly affect the eating habits and preferences of individuals. As with all chronic diseases, it is very important for individuals who continue HD treatment to comply with the drug treatment program, diet and fluid restrictions in order to maintain their health. refers to a fast and concise presentation format. It was created in 2003 by architects Astrid Klein and Mark Dytham, who hoped to give young designers the opportunity to present their work in a short, fast-paced setting. In a PK presentation, each presenter is only allowed to show 20 PowerPoint slides for 20 seconds each on a timer. In other words, the presenter has only 20 seconds to discuss each slide before the next slide appears, and the presentation time is limited to 6 minutes and 40 seconds. Ideas are explained visually with pictures and graphics, and there is little text on the slides.

ELIGIBILITY:
Inclusion Criteria:

* The patient does not have any impairment (such as vision, speech and hearing) that prevents him from communicating.
* Accepting the research
* Being receiving hemodialysis treatment
* Ability to communicate adequately
* Absence of psychiatric problems

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-28 (Estimated)

PRIMARY OUTCOMES:
Attitude Scale Towards Dietary Treatment of Hemodialysis Patients | 1 hours later
  "Attitude Scale Towards Dietary Treatment of Hemodialysis Patients" is a 16-item scale developed by Onbe and Kanda in 2018 to determine the attitudes of patients towards diet therapy. It is a 4 likert scale.
  Each item represents 1-Strongly agree, 2-Agree, 3-Disagree, 4-Strongly Disagree. This scale consists of 3 sub-dimensions.
  1. Sub size; "Behavioral tendency affected by cognition" includes 7 items (1,2,3,4,5,6,7).
  2. Sub-dimension; "Behavioral tendency affected by food culture" includes 6 (8,9,10,11,12,13) items.
  3. Sub-dimension; "Negative effect that changes diet" includes 3 items (14,15,16). The last three items in the scale are reversed.
  Higher scores obtained from the scale indicate that attitudes are better. Effect on Retention and Fluid Restriction Compliance
Dialysis Diet and Fluid Restriction Compliance Scale | 1 hours later
  It was developed by Vlaminck et al. (2001), and its Turkish validity and reliability study was performed by Kara (2009) in hemodialysis patients. WHO is a four-item self-report tool used to evaluate non-adherence to diet and fluid intake restriction in hemodialysis patients. Two items in the scale deal with diet (items 1 and 2), and the other two deal with fluid restriction (items 3 and 4) in terms of frequency and degree. The frequency of non-compliance with diet and fluid restriction is based on the behaviors of the patients in the previous 14 days. The degree of non-compliance with diet and fluid restriction has a Likert-type structure scored between 0-4 (No non-compliance = 0, Mild = 1, Moderate = 2, Severe = 3, Very severe =4) The Cronbach alpha coefficient of the scale was reported as 0.70.

CONTACTS AND LOCATIONS:
Locations (1):
- Gülcan B Turan, Elâzığ, Merkez, Turkey (Türkiye)